CLINICAL TRIAL: NCT01218334
Title: A Randomized, Single Blind, Comparative Trial of Standardized 12 Lead ECG to the 12 Lead ECG Glove for the Assessmant of Cardiac Electrical Function
Brief Title: A Comparative Trial of Standard 12 Lead ECG to the 12 Lead ECG Glove to Assess Cardiac Electrical Function
Acronym: HandEKG
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06-777
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Electrical Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Cardiac Inpatient
- 2: Cardiac Outpatient
- 3: Cardiac Clinic Patient
  Interventions: Device: 12 Lead Glove

INTERVENTIONS:
Device: 12 Lead Glove — Comparison of EKG's derived from the 12 Lead Glove vs. the Gold Standard EKG machine
  Groups: 3

SUMMARY:
The proposed study is a two-arm, randomized, single-blinded, cross-over Phase III clinical trial in which patients in 3 distinct clinical scenarios will receive the 12LEG, followed by the standard ECG, or vice-versa. Each participant will then apply the Hand ECG themselves. The 3 clinical scenarios will be: 1. patients at preoperative assessment for elective cardiac catheterization or electrophysiology procedures; 2. patients coming for outpatient cardiology appointments; 3. Inpatients admitted with a cardiac diagnosis.

The electrophysiologists reviewing ECGs will be blinded to the equipment utilized to obtain the ECG.

ELIGIBILITY:
Inclusion Criteria:

1. Preop assessment for elective cardiac catheterization or EP procedure.
2. Outpatient cardiology appointments.
3. Inpatients admitted with a cardiac diagnosis

Exclusion Criteria:

1. Age less than 18.
2. Skin breakdown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology Patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
comparison of Hand ECG to standard ECG with physician over-read | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Aizer, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States